CLINICAL TRIAL: NCT03658278
Title: Improving Preoperative Screening and Postoperative Nutrition in Trauma Patients: Does it Decrease Muscle Wasting or Complications
Brief Title: Trauma Screening and Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael C Willey (Other)
Collaborators: Orthopaedic Trauma Association (Other)
Responsible Party: Sponsor-Investigator, Michael C Willey, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201706789
Record Dates: First submitted 2018-08-31; First posted 2018-09-05 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Trauma; Nutritional Deficiency; Wound Heal
MeSH Terms: conditions — Wounds and Injuries; Malnutrition

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional supplement group (Experimental): Subjects in this group will be asked to consume the nutritional supplement on a daily basis, in addition to standard nutrition. Subjects will have pain medication and postoperative therapies per standard of care.
  Interventions: Dietary Supplement: Juven
- Standard nutrition group (No Intervention): Subjects in this group will have standard nutrition provided per dietitian recommendation. Subjects will have pain medication and postoperative therapies per standard of care.

INTERVENTIONS:
Dietary Supplement: Juven — Nutritional supplement (Juven) will be consumed daily per manufacturer recommendations
  Arms: Nutritional supplement group

SUMMARY:
The purpose of the proposed study is twofold: 1) The investigators will evaluate ultrasound imaging to screen trauma patients to identify patients at increased risk of postoperative complications associated with sarcopenia. 2) The investigators will evaluate a commercially-available oral nutritional supplement that has previously been evaluated in critically-ill intensive care patients and shown benefit for decreasing complications including decreased wound healing complications, decreased pressure ulcers, decreased skeletal muscle loss due to immobilization, and decreased one-year mortality.

DETAILED DESCRIPTION:
Following consent, patients will be assigned a unique study identification number (ID). A master list linking patient ID to patient name and medical record number will be maintained on a password protected and encrypted departmental server location with access limited to research staff. Patients will be randomized by the research team using Microsoft Word random number generator. Patients will not be blinded to their research group, as the experimental nutrition supplementation group will be asked to consume the nutritional supplement daily for a period of two weeks following surgery.

Following consent, the patient's medical record will be reviewed to identify any condition meeting exclusion criteria. If patient meets inclusion criteria we will obtain the following data to be recorded in the research database.

1. Age
2. Sex
3. Height
4. Weight
5. BMI
6. medical comorbidities necessary to calculate Charlson Comorbidity Index (myocardial infarction, congestive heart failure, peripheral vascular disease, cerebrovascular disease, dementia, chronic pulmonary disease, rheumatologic disorder, peptic ulcer disease, diabetes without chronic complications, diabetes with chronic complications, hemiplegia or paraplegia, renal disease, any malignancy, metastatic solid tumor, mild liver disease, moderate or severe liver disease, HIV/AIDS
7. MSSA (methicillin-susceptible Staphylococcus aureus) /MRSA (methicillin-resistant Staphylococcus aureus) nasal colonization status (standard preoperative evaluation)
8. tobacco use history
9. history of DVT (deep vein thrombosis) or PE (pulmonary embolism)
10. other injuries associated with current trauma to calculate Injury Severity Score

Patients will be treated with operative fixation of their fracture per standard of care. Within 24 hours of providing informed consent, we will obtain patient weight with a clinical scale or hospital bed equipped with clinical scale. We will obtain body composition using a validated handheld ultrasound device that reports fat mass, fat free mass, and % body fat (BodyMetrix, Intellimatrix, Brentwood, CA). Hand grip strength will be assessed with the patient's dominant hand, or non-dominant hand if unable to perform due to injury (hand dynamometer, Hausmann Industries, Northvale, New Jersey).

Following surgery, patients in the treatment group will be asked to consume the nutritional supplement on a daily basis, in addition to standard nutrition. The control group will have standard nutrition provided per dietitian recommendation. Patients will have pain medication and postoperative therapies per standard of care.

The nutritional supplements will be consumed per manufacturer recommendations. Descriptions of nutritional supplementation are included below.

Juven is an oral nutritional supplement produced by Abbot Nutrition. It is not considered a drug and is not under FDA regulation. Juven has been studied in clinical trials and shown to decrease pressure ulcer occurrence, decrease muscle wasting, and increase collagen deposition in wound healing (10,11).

Juven is packaged as a powder containing 24g per pouch and is mixed with 8-10 fl oz water or juice for consumption. The recommended supplementation schedule is two servings daily in addition to balanced diet.

Nutrient data for Juven obtained from manufacturer's website 7/20/2017: https://abbottnutrition.com/juven Serving size: 24 g (1 packet) L-arginine 7g L-glutamine 7g Carbohydrate 7.9g Sugars 1g Calcium 200mg Calcium beta-hydroxy-beta-methylbutyrate 1.5g

After discharge from the hospital, we will communicate with patients by mobile phone messaging on a daily basis to confirm consumption of the investigative nutritional supplementation. We will also communicate with patients at 3 months, 6 months, 9 months, and 12 months after surgery to inquire about any complications or hospitalizations.

Following surgery, patients will be reevaluated in the orthopedic trauma clinic at routine intervals per standard of care (postoperative visits are typically scheduled at 2 weeks, 6 weeks, 6 months, and 1 year). Patients will be seen in clinic by orthopedic surgery trauma staff. All orthopedic trauma staff are included on the research team. As part of routine clinical follow up visit, research team will review the patient medical record, perform a focused history and physical exam and document any new hospital readmission, medical complication, surgical complication. Radiographs will be obtained per standard orthopedic care to assess fracture healing and no additional radiographs will be obtained for the purpose of this study.

At the patient's first postoperative clinic follow up, we will repeat measures of patient weight, body composition, and hand grip strength. These measures are expected to take less than 15 minutes at the time of their clinic appointment.

Subjects will also be asked to complete several questionnaires via RedCap at several times points during the study. The questionnaires will be completed either in clinic on a tablet or computer, or a secure link to the study will be emailed to subjects.

No data collection is planned after one year from the time of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute fracture of the upper extremity, pelvis, or lower extremity with plans for operative fixation

Exclusion Criteria:

* Patients with comorbidities excluding the use of proposed nutritional supplement (phenylketonuria, galactoseria)
* Patients with major head trauma
* Pregnant women

Dementia

Vulnerable populations (minors, prisoners)

Lack of decision making capacity

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
Change in body composition | One year
  Change in muscle mass

SECONDARY OUTCOMES:
Change in hand grip strength | One year
  Change in hand grip strength as measured by hand held dynamometer
Number of participants with post-operative complications | One year
  Medical and surgical complications following operative fracture fixation, validated patient reported outcome measures, radiographic measures of fracture healing, time spent in hospital, discharge status (home versus acute rehabilitation versus skilled nursing facility)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Hendrickson, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No